CLINICAL TRIAL: NCT03332472
Title: Evaluation of Telemedicine on Metabolic Control in the Care of Diabetes Mellitus Type 1 Patients in Multiple Doses of Insulin Treatment in Andalusian Community
Brief Title: Telemedicine on Metabolic Control in Type 1 Diabetes Mellitus Andalusian Patients (PLATEDIAN)
Acronym: PLATEDIAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Andaluza de Endocrinología, Diabetes y Nutrición (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLATEDIAN
Record Dates: First submitted 2017-07-24; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Telemedicine
Keywords: type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemedicine group (Experimental): Telematics visit in front of the conventional visit face to face
  Interventions: Other: Telemedicine group
- Conventional group (Placebo Comparator): Group with conventional medical visit
  Interventions: Other: Conventional group

INTERVENTIONS:
Other: Telemedicine group
  Arms: Telemedicine group
Other: Conventional group
  Arms: Conventional group

SUMMARY:
To assess the effect of a 6-month telemedicine program (DiabeTIC) in patients with type 1 diabetes mellitus (DM1) and regular metabolic control (HbA1c <8%) in multi-dose insulin treatment (MDI) measured HbA1c vs. conventional medical care.

DETAILED DESCRIPTION:
The substitution of face-to-face visits for telematics visits has a similar effect on glycemic control (measured by HbA1c) in patients with DM1 treated with multiple daily doses of insulin (MDI) and regular metabolic control (HbA1c <8 %). It even saves costs and consumption of health resources, and improves the quality of life and satisfaction of subjects with DM1

To evaluate the effect of a 6-month Diabetic platform on telemedicine in patients with DM1 and regular metabolic control (HbA1c <8%) on MDI treatment in the following parameters:

A) Glycemic control: Mean glycemia, number of mild hypoglycemia / week, number of severe hypoglycemia / 6 months, number of hyperglycemia greater than 250mg / dl / week, number of episodes of ketosis / 6 months, number of episodes of ketoacidosis / 6meses , Number of hospital admissions due to glycemic decompensation / 6 months.

B) Glycemic variability: Standard deviation, mean amplitude of glycemic excursions (MAGE).

C) Fear of hypoglycemia: scale FH-15. D) Quality of life: Diabetes Quality of Life Questionnaire (DQoL). E) Stress: DDS questionnaire.

F) Costs and consumption of health resources:

-Cost-effectiveness (HbA1C)

ELIGIBILITY:
Inclusion Criteria:

* Patients with DM1 over 2 years of evolution.
* Age ≥18 and <65 years.
* HbA1c prior to inclusion of the study <8% (the measure being valid in the month prior to inclusion in the study)
* Intensive insulin therapy with basal-bolus MDI.
* Patients living in Andalusian
* Patients candidates for telemonitoring.
* Patients who have received written informed consent.

Exclusion Criteria:

* Treatment with ISCI.
* Chronic kidney disease, liver disease, thyroid dysfunction (except hypothyroidism correctly treated and controlled).
* Pregnancy or pregnancy planning.
* Diabetes mellitus type 2.
* Severe psychological disturbances.
* Absence of collaboration (informed consent).
* Patients who are participating in other clinical studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months
  Glycosylated hemoglobin

SECONDARY OUTCOMES:
Total daily dose of insulin | 6 months
  total daily doseof insulin (IU/day)
Total daily dose of insulin by weight | 6 months
  Total daily dose by weight (IU / kg / day)
Number of mild hypoglycaemia | 6 months
  Acude complications prior to V1: number of mild hypoglycaemia
Number of severe hypoglycemia | 6 months
  Acute complications prior to V1: number of severe hypoglycemia
Number of hyperglycemia greater than 250 mg / dl / week | 6 months
  Acute complications prior to V1: number of hyperglycemia greater than 250 mg / dl / week
Number of episodes of ketosis number of episodes of ketoacidosis | 6 months
  Acute complications prior to V1: number of episodes of ketosis and number of episodes of ketoacidosis
Number of hospital admissions due to glycemic decompensations | 6 months
  Acute complications prior to V1:number of hospital admissions due to glycemic decompensations.
Fear of hypoglycemia: FH-15 scale | 6 months
  Hypoglycemia Fear test: FH-15 questionnaire (Annex)
Quality of life | 6 months
  Diabetes Quality of Life Questionnaire (DQoL).
Stress: DDS questionnaire | 6 months
  Diabetes Distress Scale (DDS) (Polonski et al, 2005)
Time invested in the care of each patient | 6 months
  Costs and consumption of health resources: Time invested in the care of each patient in minutes
Number of telephone calls | 6 months
  Costs and consumption of health resources: Number of telephone calls
Number of face-to-face visits | 6 months
  Costs and consumption of health resources: Number of face-to-face visits
Analytics performed in the center | 6 months
  Costs and consumption of health resources: Analytics performed in the center
Analytic done in domestic scope with glucometer | 6 months
  Costs and consumption of health resources:Number of analytic done in domestic scope with glucometer
Cost of hypoglycaemic treatment (insulin) | 6 months
  Costs and consumption of health resources: Cost in of hypoglycaemic treatment (insulin) in euros.
Costs and consumption of health resources | 6 months
  Costs and consumption of health resources: Cost of number of admissions in emergencies and number of hospitalizations
Costs associated with the time spent going to the patient's hospital and family members | 6 months
  Costs and consumption of health resources: costs associated with the time spent going to the patient's hospital and family members
Costs associated with days lost due to complications. | 6 months
  Costs and consumption of health resources: costs associated with days lost due to complications.
Mean blood glucose | 6 months
  Glycemic control: Mean blood glucose (mg / dL)
Standard deviation | 6 months
  Glycemic control: Standard deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional Universitario de Málaga. Unidad de Diabetes, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Effect of intensive diabetes treatment on the development and progression of long-term complications in adolescents with insulin-dependent diabetes mellitus: Diabetes Control and Complications Trial. Diabetes Control and Complications Trial Research Group. J Pediatr. 1994 Aug;125(2):177-88. doi: 10.1016/s0022-3476(94)70190-3. PMID 8040759
- [Background] American Diabetes Association. Standards of medical care in diabetes--2012. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S11-63. doi: 10.2337/dc12-s011. No abstract available. PMID 22187469
- [Background] Chase HP, Pearson JA, Wightman C, Roberts MD, Oderberg AD, Garg SK. Modem transmission of glucose values reduces the costs and need for clinic visits. Diabetes Care. 2003 May;26(5):1475-9. doi: 10.2337/diacare.26.5.1475. PMID 12716807
- [Background] Biermann E, Dietrich W, Standl E. Telecare of diabetic patients with intensified insulin therapy. A randomized clinical trial. Stud Health Technol Inform. 2000;77:327-32. PMID 11187566
- [Background] Charpentier G, Benhamou PY, Dardari D, Clergeot A, Franc S, Schaepelynck-Belicar P, Catargi B, Melki V, Chaillous L, Farret A, Bosson JL, Penfornis A; TeleDiab Study Group. The Diabeo software enabling individualized insulin dose adjustments combined with telemedicine support improves HbA1c in poorly controlled type 1 diabetic patients: a 6-month, randomized, open-label, parallel-group, multicenter trial (TeleDiab 1 Study). Diabetes Care. 2011 Mar;34(3):533-9. doi: 10.2337/dc10-1259. Epub 2011 Jan 25. PMID 21266648
- [Background] Franc S, Daoudi A, Mounier S, Boucherie B, Dardari D, Laroye H, Neraud B, Requeda E, Canipel L, Charpentier G. Telemedicine and diabetes: achievements and prospects. Diabetes Metab. 2011 Dec;37(6):463-76. doi: 10.1016/j.diabet.2011.06.006. Epub 2011 Sep 1. PMID 21889388
- [Background] Benhamou PY, Melki V, Boizel R, Perreal F, Quesada JL, Bessieres-Lacombe S, Bosson JL, Halimi S, Hanaire H. One-year efficacy and safety of Web-based follow-up using cellular phone in type 1 diabetic patients under insulin pump therapy: the PumpNet study. Diabetes Metab. 2007 Jun;33(3):220-6. doi: 10.1016/j.diabet.2007.01.002. Epub 2007 Mar 28. PMID 17395516
- [Background] Gomez EJ, Hernando ME, Garcia A, Del Pozo F, Cermeno J, Corcoy R, Brugues E, De Leiva A. Telemedicine as a tool for intensive management of diabetes: the DIABTel experience. Comput Methods Programs Biomed. 2002 Aug;69(2):163-77. doi: 10.1016/s0169-2607(02)00039-1. PMID 12100795
- [Background] Rigla M, Hernando ME, Gomez EJ, Brugues E, Garcia-Saez G, Torralba V, Prados A, Erdozain L, Vilaverde J, de Leiva A. A telemedicine system that includes a personal assistant improves glycemic control in pump-treated patients with type 1 diabetes. J Diabetes Sci Technol. 2007 Jul;1(4):505-10. doi: 10.1177/193229680700100408. PMID 19885113
- [Background] Bellazzi R, Larizza C, Montani S, Riva A, Stefanelli M, d'Annunzio G, Lorini R, Gomez EJ, Hernando E, Brugues E, Cermeno J, Corcoy R, de Leiva A, Cobelli C, Nucci G, Del Prato S, Maran A, Kilkki E, Tuominen J. A telemedicine support for diabetes management: the T-IDDM project. Comput Methods Programs Biomed. 2002 Aug;69(2):147-61. doi: 10.1016/s0169-2607(02)00038-x. PMID 12100794
- [Background] Farmer AJ, Gibson OJ, Dudley C, Bryden K, Hayton PM, Tarassenko L, Neil A. A randomized controlled trial of the effect of real-time telemedicine support on glycemic control in young adults with type 1 diabetes (ISRCTN 46889446). Diabetes Care. 2005 Nov;28(11):2697-702. doi: 10.2337/diacare.28.11.2697. PMID 16249542
- [Background] Jansa M, Vidal M, Viaplana J, Levy I, Conget I, Gomis R, Esmatjes E. Telecare in a structured therapeutic education programme addressed to patients with type 1 diabetes and poor metabolic control. Diabetes Res Clin Pract. 2006 Oct;74(1):26-32. doi: 10.1016/j.diabres.2006.03.005. Epub 2006 Apr 18. PMID 16621113
- [Background] Montori VM, Helgemoe PK, Guyatt GH, Dean DS, Leung TW, Smith SA, Kudva YC. Telecare for patients with type 1 diabetes and inadequate glycemic control: a randomized controlled trial and meta-analysis. Diabetes Care. 2004 May;27(5):1088-94. doi: 10.2337/diacare.27.5.1088. PMID 15111526
- [Background] Rossi MC, Nicolucci A, Di Bartolo P, Bruttomesso D, Girelli A, Ampudia FJ, Kerr D, Ceriello A, Mayor Cde L, Pellegrini F, Horwitz D, Vespasiani G. Diabetes Interactive Diary: a new telemedicine system enabling flexible diet and insulin therapy while improving quality of life: an open-label, international, multicenter, randomized study. Diabetes Care. 2010 Jan;33(1):109-15. doi: 10.2337/dc09-1327. Epub 2009 Oct 6. PMID 19808926
- [Background] Anarte Ortiz MT, Caballero FF, Ruiz de Adana MS, Rondan RM, Carreira M, Dominguez-Lopez M, Machado A, Gonzalo-Marin M, Tapia MJ, Valdes S, Gonzalez-Romero S, Soriguer FC. Development of a new fear of hypoglycemia scale: FH-15. Psychol Assess. 2011 Jun;23(2):398-405. doi: 10.1037/a0021927. PMID 21381839
- [Derived] Ruiz de Adana MS, Alhambra-Exposito MR, Munoz-Garach A, Gonzalez-Molero I, Colomo N, Torres-Barea I, Aguilar-Diosdado M, Carral F, Serrano M, Martinez-Brocca MA, Duran A, Palomares R; Diabetes Group of SAEDYN (Andalusian Society of Endocrinology, Diabetes, and Nutrition). Randomized Study to Evaluate the Impact of Telemedicine Care in Patients With Type 1 Diabetes With Multiple Doses of Insulin and Suboptimal HbA1c in Andalusia (Spain): PLATEDIAN Study. Diabetes Care. 2020 Feb;43(2):337-342. doi: 10.2337/dc19-0739. Epub 2019 Dec 12. PMID 31831473